CLINICAL TRIAL: NCT00644566
Title: Pilot Study of Shared Care of ADHD in a Pediatric Clinic:Colocation of a Psychologist as an ADHD Care Manager
Acronym: shared care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); New York State Psychiatric Institute (Other); Research Foundation for Mental Hygiene, Inc. (Other); Columbia University (Other)
Responsible Party: Daniel Hyman, M.D., M.M.M., New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0604008460
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: ADHD
Keywords: ADHD; Primary Care; Pediatrics; Health services; shared care; care manager; screening
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

ARMS (2):
- TAU (No Intervention): Treatment as usual. These subjects and their providers were told to pursue treatment services as they normally would do.
- shared care (Experimental): A psychologist co-located in the pediatric primary care clinic shared care with the subject's pediatrician. The psychologist offered regular appointments and psychoeducation. On an individual basis, parent management training, behavioral management training, individual psychotherapy, educational intervention assistance, teacher communication, and medication education were provided as needed.
  Interventions: Other: Shared Care

INTERVENTIONS:
Other: Shared Care — A psychologist co-located in the pediatric primary care clinic shared care with the subject's pediatrician. The psychologist offered regular appointments and psychoeducation. On an individual basis, parent management training, behavioral management training, individual psychotherapy, educational intervention assistance, teacher communication, and medication education were provided as needed.
  Arms: shared care

SUMMARY:
Due to the shortage of child psychiatrists and the high prevalence of child mental health disorder, pediatricians and other pediatric primary care providers often assume responsibility for the management of various psychiatric disorders, including ADHD, Attention Deficit Hyperactivity Disorder. However, pediatricians have not been well-trained during residency to deal with the complexities of ADHD management. In addition, the system of care under which pediatricians practice do not afford the time availability that is required to properly manage a child with ADHD. On the other hand, if a pediatrician wishes to refer a patient to a child mental health specialist, many obstacles, including but not limited to stigma, insurance issues, and long waiting lists, often interfere with the patient actually receiving services for his/her ADHD. This research project seeks to examine an innovative model of care in which a child psychologist is located on the premises of a pediatric office and is available to share the care of patients with the pediatrician in order to address ADHD. We hypothesize that parents as well as pediatricians will be more satisfied with this model of care and that patients will ultimately have better outcomes. The beginning of our pilot has shown under-identification to be a barrier to care as well, and thus we propose to implement a quality improvement initiative to screen children for psychosocial issues as well. As we have had trouble with recruitment and unfortunately have had more children randomized to TAU than shared care, we propose in December 2007 a phase 2 of our study where all subjects, instead of randomization, are entered into shared care.

DETAILED DESCRIPTION:
Study Goals:

A. To compare patients with ADHD (Attention Deficit Hyperactivity Disorder) treated by a pediatric provider in collaboration with a co-located psychologist/ADHD care manager available for evaluation/assessment and ongoing shared-care consultation to patients with ADHD in a pediatric primary care clinic treated as usual.

1. Patients treated by the pediatricians with the added co-located services will have clinical outcomes that are superior to those that receive usual care

   1. Co-located services will increase the number of ADHD patients accessing specialized mental health treatment services
   2. A higher proportion of patients treated by the pediatric providers and psychologists than those in usual care receive doses of medication that are consistent with AAP (American Academy of Pediatrics) recommendations
2. Patients whose providers are offered to receive the aid of the co-located psychologists will be more likely to be co-managed by the pediatrician than referred out to the community.
3. Parents will be more satisfied with care in the shared care model than in usual care

B. Pediatricians' morale and attitudes to the treatment of ADHD will improve with the addition of a co-located psychologist.

C. ADDITIONAL AIMS:

1. To assist a pediatric primary care clinic in implementing a quality improvement initiative to help pediatric providers better identify ADHD by implementing the PSC-17, a general psychosocial checklist.
2. Study the usefulness of using the PSC 17 screen as a clinical tool to identify ADHD in the primary care office by obtaining results and tracking physician disposition planning based on results.

D. Operationalize Shared Care by examining what happens in such an arrangement, and see if patient recruitment and provider buy-in improves when shared care is assured.

ELIGIBILITY:
Inclusion Criteria (Patient subjects):

* Age 6-17
* Suspected diagnosis of ADHD, inattentive type, hyperactive type, combined type, NOS
* Living with Guardian for at least 6 months
* English-speaking child
* English-speaking guardian
* Telephone Access to Guardian
* Inclusion for Randomization or Phase 2 shared care:
* Diagnosis of ADHD

Exclusion Criteria:

* Mental Retardation
* Co-morbid psychotic disorder
* Suicidal
* Homicidal
* Dangerous behavior
* Foster care
* Impairing co-morbid psychiatric disorder that would make ADHD treatment in a pediatric clinic unsafe or inappropriate (in the judgment of the PI based on the case review of the findings of the clinical psychologist.)
* Allergic or contraindication to stimulant medications

Inclusion Criteria (Provider subjects):

* Provider at Cornell Campus Helmsley Tower 5/ Long Island City Campus

Exclusion Criteria:

* None

Inclusion for screening:

* Age 6-17
* Child is to be seen by pediatric provider at HT5
* Parent or guardian reads English or Spanish

Exclusion Criteria:

* Parent/Guardian has received screen within the year
* Patient is too sick for parent to spend time on form

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
A higher proportion of patients treated by the pediatric providers and psychologists than those in usual care receive doses of medication that are consistent with AAP (American Academy of Pediatrics) recommendations | six months

SECONDARY OUTCOMES:
Co-located services will increase the number of ADHD patients accessing specialized mental health treatment services | six months
2. Patients whose providers are offered to receive the aid of the co-located psychologists will be more likely to be co-managed by the pediatrician than referred out to the community. | six months
Parents will be more satisfied with care in the shared care model than in usual care | six months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hyman, MD, Principal Investigator — New York Presbyterian Hospital; Rachel Zuckerbrot, MD, Principal Investigator — Columbia University/New York State Psychiatric Institute; Mark Olfson, MD, Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Long Island City Community Practice, Long Island City, New York
  - New York Presbyterina Hospital- Weill Cornell Medcial College HT5 Pediatrics Clinic, New York, New York